CLINICAL TRIAL: NCT04197479
Title: A 52-Week, Phase 3 Study to Evaluate Safety and Biomarkers of Resmetirom (MGL-3196) in Patients With Non-alcoholic Fatty Liver Disease (NAFLD) (MAESTRO-NAFLD-1)
Brief Title: A Phase 3 Study to Evaluate Safety and Biomarkers of Resmetirom (MGL-3196) in Non Alcoholic Fatty Liver Disease Patients
Acronym: MAESTRO-NAFLD1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Madrigal Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MGL-3196-14
Record Dates: First submitted 2019-12-11; First posted 2019-12-13 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2023-08

CONDITIONS: Non-Alcoholic Fatty Liver Disease
Keywords: NAFLD; NASH; Hyperlipidemia; Resmetirom; Thyroid hormone receptor beta; Hepatic; Fibrosis; NASH resolution; Thyroid hormone receptor agonist; Cardiovascular; Dyslipidemia; Fatty liver disease; Nonalcoholic steatohepatitis; Cirrhosis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Hyperlipidemias; Thyroid Hormone Resistance Syndrome; Fibrosis; Dyslipidemias | interventions — resmetirom

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Open label: resmetirom (Experimental): 100 mg daily
  Interventions: Drug: Resmetirom
- Double blinded: matching placebo (Placebo Comparator): Placebo daily
  Interventions: Drug: Placebo
- Double blinded: resmetirom 80 mg (Experimental): 80 mg daily
  Interventions: Drug: Resmetirom
- Double blinded: resmetirom 100 mg (Experimental): 100 mg daily
  Interventions: Drug: Resmetirom

INTERVENTIONS:
Drug: Placebo — Matching tablets
  Arms: Double blinded: matching placebo
Drug: Resmetirom — Tablet
  Other Names: MGL-3196
  Arms: Double blinded: resmetirom 100 mg; Double blinded: resmetirom 80 mg; Open label: resmetirom

SUMMARY:
A double-blind placebo controlled randomized Phase 3 study to evaluate the safety and tolerability of once-daily, oral administration of 80 or 100 mg resmetirom versus matching placebo. At least 100 patients will be enrolled in a 100 mg open-label arm and will include a special safety population (eg, patients with compensated NASH cirrhosis).

ELIGIBILITY:
Inclusion Criteria:

* Must be willing to participate in the study and provide written informed consent.
* Male and female adults ≥18 years of age.
* Suspected or confirmed diagnosis of NASH or NAFLD (presumed NASH):

  * Fibroscan with kPa ≥5.5 and <8.5; CAP ≥280 dB.m-1 OR
  * MRE ≥2 and <4.0; MRI-PDFF ≥8% liver fat consistent with steatosis and fibrosis stage ≥1 and <4. OR
  * Recent liver biopsy (within past 2 years) documenting NASH/NAFLD with steatosis showing one of the following:

    * NAS ≥4, steatosis ≥1, fibrosis stage 0 or F1A/1C with PRO-C3 <14
    * NAS <4, steatosis ≥1, with fibrosis stage ≤3
    * NAS ≥4, steatosis ≥1, fibrosis stage ≤3 without ballooning

      * NOTE: Since the completion of enrollment of the double-blind arms, patients meeting all other criteria who have a liver biopsy result from MGL-3196-11 with the following may be enrolled in the open-label active treatment arm of MGL-3196-14 (100 mg dose):

        * NAS = 3, steatosis 1, ballooning 1, inflammation 1 with F2 or F3
        * NAS = 3, ballooning 0 with F2 or F3
      * For the compensated NASH cirrhosis arm, eligible patients must have compensated NASH cirrhosis diagnosed by liver biopsy showing NASH with F4 stage fibrosis (either historic or recent biopsy) or a historic biopsy with NASH F2-F3 fibrosis with subsequent progression to NASH cirrhosis as diagnosed by an expert hepatologist/gastroenterologist.
  * Compensated NASH cirrhosis at screening and baseline includes

    * Child Pugh-A (score 5-6) ( may have either mild hepatic encephalopathy OR mild diuretic responsive ascites OR albumin < 3.5 and ≥ 3.2 (not any two of these, unless explained by Gilbert's Syndrome or non-hepatic causes)).
    * MELD < 12 at screening/baseline unless MELD ≥ 12 based on non-cirrhotic parameters (e.g., elevated INR due to anticoagulation, bilirubin elevation due to documented Gilbert's Syndrome, elevated creatine due to renal disease (non-hepatic)).
    * Albumin ≥ 3.2.
    * Bilirubin < 2 (unless documented Gilbert's Syndrome).
* MRI-PDFF fat fraction ≥8% obtained during the Screening Period (baseline MRI-PDFF) or a historic MRI-PDFF ≤8 weeks old at the time of randomization.
* Stable dyslipidemia therapy for ≥30 days prior to randomization.

Exclusion Criteria:

* History of significant alcohol consumption for a period of more than 3 consecutive months within 1 year prior to Screening.
* Regular use of drugs historically associated with NAFLD.
* History of bariatric surgery or intestinal bypass surgery within the 5 years prior to randomization or planned during the conduct of the study.
* Weight gain or loss ≥5% total body weight within 12 weeks prior to randomization.
* HbA1c >9.0%.
* Glucagon-like peptide 1 [GLP-1] agonist therapy or high dose vitamin E (>400 IU/day) unless stable for 24 weeks prior to biopsy.
* Presence of cirrhosis on liver biopsy defined as stage 4 fibrosis.
* Diagnosis of hepatocellular carcinoma (HCC).
* Model for End-stage Liver Disease (MELD) score ≥12, as determined at Screening, unless due to therapeutic anti coagulation or Gilbert syndrome.
* Hepatic decompensation.
* Chronic liver diseases.
* Has an active autoimmune disease.
* Serum ALT >250 U/L.
* History of biliary diversion.
* Uncontrolled hypertension (either treated or untreated).
* Active, serious medical disease with a likely life expectancy <2 years.
* Participation in an investigational new drug trial in the 60 days or 5 half-lives, whichever is longer, prior to randomization.
* Any other condition which, in the opinion of the Investigator, would impede compliance, hinder completion of the study, compromise the well-being of the patient, or interfere with the study outcomes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1343 (Actual)
Dates: Start 2019-12-16 (Actual); Primary Completion 2023-01-06 (Actual); Study Completion 2023-01-06 (Actual)

PRIMARY OUTCOMES:
The effect of once daily, oral administration of 80 or 100 mg resmetirom versus placebo on the incidence of adverse events. | 52 weeks
  The effect of once daily, oral administration of 80 or 100 mg resmetirom versus placebo on the incidence of adverse events.

SECONDARY OUTCOMES:
The effect of once daily, oral administration of 80 or 100 mg resmetirom versus placebo on the percent change in low density lipoprotein C (LDL-C) from baseline to Week 24 | 24 weeks
  The effect of once daily, oral administration of 80 or 100 mg resmetirom versus placebo on the percent change in low density lipoprotein C (LDL-C) from baseline to Week 24
The effect of once daily, oral administration of 80 or 100 mg resmetirom versus placebo on the percent change in apolipoprotein B (ApoB) from baseline to Week 24 | 24 weeks
  The effect of once daily, oral administration of 80 or 100 mg resmetirom versus placebo on the percent change in apolipoprotein B (ApoB) from baseline to Week 24
The effect of once daily, oral administration of 80 or 100 mg resmetirom versus placebo on the percent change in hepatic fat fraction as determined by MRI-PDFF from baseline to Week 16. | 16 weeks
  The effect of once daily, oral administration of 80 or 100 mg resmetirom versus placebo on the percent change in hepatic fat fraction as determined by MRI-PDFF from baseline to Week 16.
The effect of once daily, oral administration of 80 or 100 mg resmetirom versus placebo on the percent change in triglycerides (TGs) from baseline to Week 24 in patients with baseline TG > 150 mg/dL. | 24 weeks
  The effect of once daily, oral administration of 80 or 100 mg resmetirom versus placebo on the percent change in triglycerides (TGs) from baseline to Week 24 in patients with baseline TG > 150 mg/dL.
The effect of once daily, oral administration of 80 or 100 mg resmetirom versus placebo after 52 weeks on FibroScan controlled attenuation parameter (CAP) | 52 weeks
  The effect of once daily, oral administration of 80 or 100 mg resmetirom versus placebo after 52 weeks on FibroScan controlled attenuation parameter (CAP)
The change from baseline to Week 52 in FibroScan vibration controlled transient elastography (kPa) | 52 weeks
  The change from baseline to Week 52 in FibroScan vibration controlled transient elastography (VCTE) (kPa) in patients with baseline kPa >/=7.2 and a Week 52 or end of treatment FibroScan (VCTE)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Taub, MD, Study Director — Madrigal Pharmaceuticals, Inc.
Locations (77):
- United States (76):
  - Central Research Associates, Birmingham, Alabama
  - Arizona Liver Health - Chandler, Chandler, Arizona
  - East Valley Family Physicians, Chandler, Arizona
  - The Institute For Liver Health - Glendale, Glendale, Arizona
  - Arizona - Desert Clinical Research, Mesa, Arizona
  - The Institute For Liver Health - Tucson, Tucson, Arizona
  - Adobe Gastroenterology, Tucson, Arizona
  - Arkansas Gastroenterology, North Little Rock, Arkansas
  - Fresno Clinical Research Center, Fresno, California
  - National Research Institute - Huntington Park, Huntington Park, California
  - Ruane Clinical Research Group, Los Angeles, California
  - National Research Institute - Los Angeles, Los Angeles, California
  - Catalina Research Institute, Montclair, California
  - National Research Institute - Panorama City, Panorama City, California
  - Alliance Clinical Research, Poway, California
  - San Fernando Valley Health Institute, West Hills, California
  - South Denver Gastroenterology - Swedish Medical Center Office, Englewood, Colorado
  - Excel Medical Clinical Trials, Boca Raton, Florida
  - Velocity Clinical Research, Hallandale Beach (MD Clinical), Hallandale, Florida
  - Floridian Clinical Research, Hialeah, Florida
  - Nature Coast Clinical Research - Inverness, Inverness, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Florida Research Institute, Lakewood Rch, Florida
  - Miami Dade Medical Research Institute, Miami, Florida
  - Orlando Research Center, Orlando, Florida
  - Progressive Medical Research, Port Orange, Florida
  - Covenant Research, Sarasota, Florida
  - The Villages Research Center, The Villages, Florida
  - Gastrointestinal Specialists of Georgia, Marietta, Georgia
  - East-West Medical Research Institute, Honolulu, Hawaii
  - Chicago Research Center, Chicago, Illinois
  - Northwestern Memorial Physicians Group, Chicago, Illinois
  - Iowa Diabetes Research, West Des Moines, Iowa
  - Kansas Medical Clinic - Gastroenterology, Topeka, Kansas
  - L-MARC Research Center, Louisville, Kentucky
  - Digestive Health Center of Louisiana, Baton Rouge, Louisiana
  - Tandem Clinical Research - New Orleans Area Site, Marrero, Louisiana
  - Clinical Trials of America, West Monroe, Louisiana
  - Huron Gastroenterology, Ypsilanti, Michigan
  - Gastrointestinal Associates & Endoscopy Center - Flowood, Flowood, Mississippi
  - Southern Therapy and Advanced Research, Jackson, Mississippi
  - Kansas City Research Institute, Kansas City, Missouri
  - Henderson Research Center, Henderson, Nevada
  - Clarity Clinical Research, East Syracuse, New York
  - Mount Sinai Health System, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Cumberland Research Associates, Fayetteville, North Carolina
  - Diabetes and Endocrinology Consultants, Morehead City, North Carolina
  - TMA - Wilmington Gastroenterology Accociates, Wilmington, North Carolina
  - Platinum - Sterling Research Group - Springdale, Cincinnati, Ohio
  - Aventiv Research Columbus, Columbus, Ohio
  - Awasty Research Network, Marion, Ohio
  - Northeast Clinical Research Center, Bethlehem, Pennsylvania
  - Premier Medical Group - Clarksville - Dunlop Lane, Clarksville, Tennessee
  - Gastro One - Germantown Office - Wolf Park Drive, Germantown, Tennessee
  - Pinnacle Clinical Research - Austin, Austin, Texas
  - The Liver Institute At Methodist Dallas, Dallas, Texas
  - Dallas Research Center, Dallas, Texas
  - Liver Center of Texas, Dallas, Texas
  - Texas Digestive Disease Consultants - Dallas - Baylor University Medical Center Gaston Ave, Dallas, Texas
  - South Texas Research Institute, Edinburg, Texas
  - Texas Digestive Disease Consultants - Forth Worth - Downtown, Fort Worth, Texas
  - Liver Associates of Texas, Houston, Texas
  - Doctor's Hospital at Renaissance, McAllen, Texas
  - Plano Research Center, Plano, Texas
  - Texas Liver Institute/American Research Corporation, San Antonio, Texas
  - Pinnacle Clinical Research - San Antonio, San Antonio, Texas
  - San Antonio Research Center, San Antonio, Texas
  - Texas Digestive Disease Consultants - San Marcos, San Marcos, Texas
  - Texas Digestive Disease Consultants - Bay Area Houston Endoscopy Center, Webster, Texas
  - Wasatch Peak Family Practice, Layton, Utah
  - Salt Lake City Research Center, Murray, Utah
  - Bon Secours Liver Institute of Richmond, Richmond, Virginia
  - National Clinical Research - Richmond, Richmond, Virginia
  - Virginia Commonwealth University School of Medicine, Richmond, Virginia
  - Liver Institute Northwest, Seattle, Washington
- Fundacion de Investigacion de Diego, San Juan, Puerto Rico

REFERENCES:
- [Derived] Alkhouri N, McRae MP, Taub R, Hill B, Imperial JC, Kittelson J, Moussa SE, Everson GT. The Cholate Challenge Test Quantified Baseline Functional Heterogeneity and Improvement in Response to Resmetirom in MASH-related Child-Pugh A Cirrhosis. Gastro Hep Adv. 2025 Aug 29;4(10):100785. doi: 10.1016/j.gastha.2025.100785. eCollection 2025. PMID 41142528
- [Derived] Harrison SA, Taub R, Neff GW, Lucas KJ, Labriola D, Moussa SE, Alkhouri N, Bashir MR. Resmetirom for nonalcoholic fatty liver disease: a randomized, double-blind, placebo-controlled phase 3 trial. Nat Med. 2023 Nov;29(11):2919-2928. doi: 10.1038/s41591-023-02603-1. Epub 2023 Oct 16. PMID 37845512
- [Derived] Harrison SA, Ratziu V, Anstee QM, Noureddin M, Sanyal AJ, Schattenberg JM, Bedossa P, Bashir MR, Schneider D, Taub R, Bansal M, Kowdley KV, Younossi ZM, Loomba R. Design of the phase 3 MAESTRO clinical program to evaluate resmetirom for the treatment of nonalcoholic steatohepatitis. Aliment Pharmacol Ther. 2024 Jan;59(1):51-63. doi: 10.1111/apt.17734. Epub 2023 Oct 2. PMID 37786277